CLINICAL TRIAL: NCT02060058
Title: Boceprevir-based Triple Therapy to Rescue HCV Genotype 1/HBV Dually Infected Patients Refractory to Peginterferon Plus Ribavirin Combination Therapy
Brief Title: Boceprevir-based Therapy to Rescue HCV Genotype 1/HBV Infected Patients Refractory to Combination Therapy
Acronym: BOLERO-CB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-2013-10-03 (I)
Record Dates: First submitted 2014-01-27; First posted 2014-02-11 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2016-05

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C virus; hepatitis B virus; boceprevir; null responder; partial responder; relapser
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Hepatitis B | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patients with 32 week therapy (Experimental): For non-cirrhotic patients whose response of previous HCV therapy with PEG-IFN/RBV were relapse or partial response, PEG-IFN/RBV lead-in therapy is performed during 0-4 weeks, then add boceprevir from week 5 (boceprevir+ PEG-IFN/RBV). If HCV RNA is undetectable during 8-24 weeks, boceprevir+PEG-IFN/RBV triple therapy will be administered from week 5 to week 32.
  Dosage of drugs: Boceprevir 800mg tid po, PegIntron 1.5 mcg/kg im QW, and Ribavirin 800 to 1400 mg/day PO divided BID Regimen adjusted according to body weight.
  Stop trial intervention for patients with 32 week therapy: for all patients, if HCV RNA is more than 100 IU/ml at week 12 or HCV RNA is detectable at week 24, therapy will be stopped (Stop trial intervention for boceprevir, PEG-IFN and RBV for arm A).
  Interventions: Drug: Stop trial intervention for boceprevir, PEG-IFN and RBV
- Patients with 48 weeks therapy (Experimental): For non-cirrhotic patients whose response of previous HCV therapy with PEG-IFN/RBV were relapse or partial response, PEG-IFN/RBV lead-in therapy is performed during 0-4 weeks, then add boceprevir from week 5 (boceprevir+ PEG-IFN/RBV). If HCV RNA is detectable at week 8 and undetectable at week 24, boceprevir+ PEG-IFN/RBV triple therapy will be administered from week 5 to week 32, followed by additional 12 weeks of PEG-IFN/RBV therapy.
  Dosage of drugs: as Patients with 32 week therapy Stop trial intervention for patients with 48 weeks therapy: for all patients, if HCV RNA is more than 100 IU/ml at week 12 or HCV RNA is detectable at week 24, therapy will be stopped (Stop trial intervention for boceprevir, PEG-IFN and RBV for arm B).
  Interventions: Drug: Stop trial intervention for boceprevir, PEG-IFN and RBV
- Null responder or cirrhotic patients (Experimental): For null responder or cirrhotic patients, PEG-IFN/RBV lead-in therapy is performed during 0-4 weeks, then add boceprevir from week 5 to 48.
  Dosage of drugs: as Patients with 32 week therapy Stop trial intervention for for null responder or cirrhotic patients: for all patients, if HCV RNA is more than 100 IU/ml at week 12 or HCV RNA is detectable at week 24, therapy will be stopped (Stop trial intervention for boceprevir, PEG-IFN and RBV for arm C).
  Interventions: Drug: Stop trial intervention for boceprevir, PEG-IFN and RBV

INTERVENTIONS:
Drug: Stop trial intervention for boceprevir, PEG-IFN and RBV — Stop trial intervention for patients with 32 week therapy (arm A): for all patients, if HCV RNA is more than 100 IU/ml at week 12 or HCV RNA is detectable at week 24, therapy will be stopped.
  Stop trial intervention for patients with 48 weeks therapy (arm B): for all patients, if HCV RNA is more than 100 IU/ml at week 12 or HCV RNA is detectable at week 24, therapy will be stopped.
  Stop trial intervention for for null responder or cirrhotic patients: (arm C) for all patients, if HCV RNA is more than 100 IU/ml at week 12 or HCV RNA is detectable at week 24, therapy will be stopped.
  Other Names: Stop trial intervention for arm A; Stop trial intervention for arm B; Stop trial intervention for arm C

SUMMARY:
The aim of this study is to explore the efficacy and safety of boceprevir -based triple therapy to rescue HCV genotype 1 (HCV GT1)/HBV dually infected patients refractory to previous peginterferon (PEG-IFN) plus ribavirin (RBV) combination therapy.

DETAILED DESCRIPTION:
Liver disease, especially viral hepatitis, is an important public health issue, which frequent leads to liver cirrhosis, hepatocellular carcinoma (HCC) and liver-related death. Around 340 to 400 million persons are infected with hepatitis B virus (HBV) and 130 to 210 million persons are infected with hepatitis C virus (HCV) worldwide, In Taiwan, the prevalence of HBV infection is 15-20%, and the prevalence of HCV infection is 2-5% in general population. Moreover, there are some HCV-hyperendemic areas in southern Taiwan with anti-HCV prevalence rate of as high as 30-40%.

HBV/HCV dual infections is not uncommon in HBV epidemic areas, such as Southeastern Asia, with a prevalence rate of 1.1% in southern Taiwan. Recent study showed that the risk of HCC incidence is even higher among HBV/HCV co-infected persons than those with HBV or HCV mono-infection, indicating the importance of disease control in this clinical setting.

The PEG-IFN/RBV has been effective in the treatment of HCV-dominant, treatment-naïve patients with HCV/HBV dual infections. For treatment-naive HCV genotype 1 (HCV GT1)/HBV co-infected patients, 48 weeks of peginterferon (PEG-IFN) plus ribavirin (RBV) could achieve an HCV sustained virological response (SVR) rate of 72%, which was comparable to 77% for patients with HCV GT1 monoinfection. For treatment-naive HCV GT2 or GT3 /HBV co-infected patients, 24 weeks of PEG-IFN plus RBV could achieve an HCV SVR rate of 83%, which was comparable to 84% for patients with HCV GT2/3 monoinfection . Furthermore, PEG-IFN plus RBV combination therapy could enhance seroclearance of hepatitis B surface antigen (HBsAg) with an HBsAg loss rate of upto 11%. Nevertheless, there is about 30% of HCV GT1/HBV and 20% of HCV GT2 or 3/HBV co-infected patients refractory to current PEG-IFN/RBV combination therapy, which remains at high risk of HCC and liver-related death.

Boceprevir is an oral antiviral drug, which is NS3/4A protease inhibitor. Boceprevir has been approved for treating HCV GT1 infection by Food and Drug Administration (FDA) on 11 May 2011. For HCV GT1 mono-infected patients who refractory to previous PEG-IFN plus RBV combination therapy, becoprevir combined with PEG-IFN/RBV triple therapy can improve the treatment efficacy. The SVR rate of becoprevir-based triple therapy is about 3 times when compared to patients who received PEG-IFN with RBV dual therapy [14].The investigators , therefore, hypothesize that boceprevir plus PEG-IFN/RBV is effective in treating HCV GT1/HBV dually infected patients who are refractory to previous PEG-IFN/RBV combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient must be 20 years or older
* 2. Patient must have HCV GT1 infection combined with HBV infection.
* 3. Patients must be serum HCV RNA detectable, anti-HCV positive, HBsAg positive and HBeAg negative.
* 4. Patient has previously failed treatment with PEG-IFN-α 2a or 2b/RBV for minimum of 12 weeks of treatment.
* 5. Patient must have compensated liver disease consistent with CHC and/or CHB, and no other etiology. Note: patients with cirrhosis should have a liver imaging study (e.g. ultrasound, CT scan or MRI) within the preceding 6 months showing no evidence of hepatocellular carcinoma.
* 6. Patient meets all of the requirements and none of the contra-indications for treatment with PEG-IFN alpha-2b/RBV or boceprevir defined in the labels for the PEG-IFN/RBV to be used in combination with boceprevir.
* 7. Patient is able and willing to provide signed informed consent (prepared by and administered by the physician) as required by local country requirements.

Exclusion Criteria:

* 1. Mixed genotypes including HCV genotype other than genotype 1.
* 2. Patient has received boceprevir, narlaprevir, telaprevir, or any other HCV protease inhibitor treatment.
* 3. Patient has evidence of decompensated liver disease including but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy.
* 4. Patient meets any of the following exclusionary hematologic and biochemical criteria (documentation required) Hemoglobin <12 gm/dL for females and <13 gm/dL for males Neutrophils <1500/mm3 Platelets <100,000/mm3
* 5. Patient has an organ transplant other than cornea or hair.
* 6. Patient is co-infected with human immunodeficiency virus (HIV)
* 7. Patient requires or is anticipated to require any of the following prohibited medications: midazolam, pimozide, amiodarone, flecainide, propafenone, quinidine, and ergot derivatives
* 8. Patient with clinical diagnosis or evidence of substance abuse involving alcohol, intravenous drugs, inhalational psychotropics, narcotics, cocaine prescription or over-the-counter drugs.
* 9. Patient previously demonstrated clinically significant hypersensitivity or other contraindication to any component of the boceprevir formulation. This drug contains lactose. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption should not take this medicine.
* 10. Serious illness, including malignancy, active coronary artery disease or cardiac dysfunction within 24 weeks prior to study entry, that in the opinion of the site investigator may preclude completion of the treatment regimen.
* 11. Major hemoglobinopathy (e.g., thalassemia major), coagulopathy or any other cause of or tendency to hemolysis or bleeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, Professsor, Study Chair — Hepatitis Center and Hepatobiliary Division, Department of Internal Medicine, Kaohsiung Medical University Hospital, Kaohsiung, Taiwan
Locations (1):
- Hepatitis Center and Hepatobiliary Division, Department of Internal Medicine, Kaohsiung Medical University Hospital, Kaohsiung, Taiwan., Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Until now if sharing data is not decided

REFERENCES:
- [Background] Chuang WL, Chang WY, Lu SN, Lin ZY, Chen SC, Hsieh MY, Wang LY, You SL, Chen CJ. The role of hepatitis C virus in chronic hepatitis B virus infection. Gastroenterol Jpn. 1993 May;28 Suppl 5:23-7. doi: 10.1007/BF02989199. PMID 7689504
- [Background] Chen DS, Wang JT, Chen PJ, Wang TH, Sung JL. Hepatitis C virus infection in Taiwan. Gastroenterol Jpn. 1991 Jul;26 Suppl 3:164-6. doi: 10.1007/BF02779290. PMID 1909259
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of hepatitis C virus infection. J Hepatol. 2011 Aug;55(2):245-64. doi: 10.1016/j.jhep.2011.02.023. Epub 2011 Mar 1. No abstract available. PMID 21371579
- [Background] Papatheodoridis GV, Manolakopoulos S, Liaw YF, Lok A. Follow-up and indications for liver biopsy in HBeAg-negative chronic hepatitis B virus infection with persistently normal ALT: a systematic review. J Hepatol. 2012 Jul;57(1):196-202. doi: 10.1016/j.jhep.2011.11.030. Epub 2012 Mar 23. PMID 22450396
- [Background] Chen DS, Sung JL. Studies on the subtypes of hepatitis B surface antigen-demonstration of vertical and intrafamilial transmission of hepatitis B virus. Taiwan Yi Xue Hui Za Zhi. 1978 Mar;77(3):263-71. No abstract available. PMID 275454
- [Background] Stevens CE, Beasley RP, Tsui J, Lee WC. Vertical transmission of hepatitis B antigen in Taiwan. N Engl J Med. 1975 Apr 10;292(15):771-4. doi: 10.1056/NEJM197504102921503. PMID 1113797
- [Background] Sheu JC, Wang JT, Wang TH, Wang CY, Yang PM, Huang GT, Shih LN, Lee HS, Chen DS. Prevalence of hepatitis C viral infection in a community in Taiwan. Detection by synthetic peptide-based assay and polymerase chain reaction. J Hepatol. 1993 Feb;17(2):192-8. doi: 10.1016/s0168-8278(05)80037-6. PMID 8383160
- [Background] Yang JF, Lin CI, Huang JF, Dai CY, Lin WY, Ho CK, Hsieh MY, Lee LP, Ho NJ, Lin ZY, Chen SC, Hsieh MY, Wang LY, Yu ML, Chuang WL, Chang WY. Viral hepatitis infections in southern Taiwan: a multicenter community-based study. Kaohsiung J Med Sci. 2010 Sep;26(9):461-9. doi: 10.1016/S1607-551X(10)70073-5. PMID 20837342
- [Background] Liu CJ, Chen PJ, Chen DS. Dual chronic hepatitis B virus and hepatitis C virus infection. Hepatol Int. 2009 Dec;3(4):517-25. doi: 10.1007/s12072-009-9147-9. Epub 2009 Aug 8. PMID 19669238
- [Background] Huang YT, Jen CL, Yang HI, Lee MH, Su J, Lu SN, Iloeje UH, Chen CJ. Lifetime risk and sex difference of hepatocellular carcinoma among patients with chronic hepatitis B and C. J Clin Oncol. 2011 Sep 20;29(27):3643-50. doi: 10.1200/JCO.2011.36.2335. Epub 2011 Aug 22. PMID 21859997
- [Background] Liu CJ, Chuang WL, Lee CM, Yu ML, Lu SN, Wu SS, Liao LY, Chen CL, Kuo HT, Chao YC, Tung SY, Yang SS, Kao JH, Liu CH, Su WW, Lin CL, Jeng YM, Chen PJ, Chen DS. Peginterferon alfa-2a plus ribavirin for the treatment of dual chronic infection with hepatitis B and C viruses. Gastroenterology. 2009 Feb;136(2):496-504.e3. doi: 10.1053/j.gastro.2008.10.049. Epub 2008 Oct 29. PMID 19084016
- [Background] Potthoff A, Wedemeyer H, Boecher WO, Berg T, Zeuzem S, Arnold J, Spengler U, Gruengreiff K, Kaeser T, Schuchmann M, Bergk A, Forestier N, Deterding K, Manns MP, Trautwein C; Hep-Net B/C Co-infection Study Group. The HEP-NET B/C co-infection trial: A prospective multicenter study to investigate the efficacy of pegylated interferon-alpha2b and ribavirin in patients with HBV/HCV co-infection. J Hepatol. 2008 Nov;49(5):688-94. doi: 10.1016/j.jhep.2008.03.028. Epub 2008 Apr 29. PMID 18490077
- [Background] Yu JW, Sun LJ, Zhao YH, Kang P, Gao J, Li SC. Analysis of the efficacy of treatment with peginterferon alpha-2a and ribavirin in patients coinfected with hepatitis B virus and hepatitis C virus. Liver Int. 2009 Nov;29(10):1485-93. doi: 10.1111/j.1478-3231.2009.02080.x. Epub 2009 Jul 7. PMID 19602134
- [Background] Bacon BR, Gordon SC, Lawitz E, Marcellin P, Vierling JM, Zeuzem S, Poordad F, Goodman ZD, Sings HL, Boparai N, Burroughs M, Brass CA, Albrecht JK, Esteban R; HCV RESPOND-2 Investigators. Boceprevir for previously treated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1207-17. doi: 10.1056/NEJMoa1009482. PMID 21449784
- [Background] Zeuzem S, Andreone P, Pol S, Lawitz E, Diago M, Roberts S, Focaccia R, Younossi Z, Foster GR, Horban A, Ferenci P, Nevens F, Mullhaupt B, Pockros P, Terg R, Shouval D, van Hoek B, Weiland O, Van Heeswijk R, De Meyer S, Luo D, Boogaerts G, Polo R, Picchio G, Beumont M; REALIZE Study Team. Telaprevir for retreatment of HCV infection. N Engl J Med. 2011 Jun 23;364(25):2417-28. doi: 10.1056/NEJMoa1013086. PMID 21696308
- [Background] Yu ML, Lee CM, Chen CL, Chuang WL, Lu SN, Liu CH, Wu SS, Liao LY, Kuo HT, Chao YC, Tung SY, Yang SS, Kao JH, Su WW, Lin CL, Yang HC, Chen PJ, Chen DS, Liu CJ; Taiwan Liver-Net Consortium. Sustained hepatitis C virus clearance and increased hepatitis B surface antigen seroclearance in patients with dual chronic hepatitis C and B during posttreatment follow-up. Hepatology. 2013 Jun;57(6):2135-42. doi: 10.1002/hep.26266. Epub 2013 Apr 26. PMID 23322699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As protocol
Pre-assignment Details: As protocol
Groups:
- Patients With 32 Week Therapy: For non-cirrhotic patients whose response of previous HCV therapy with PEG-IFN/RBV were relapse or partial response, PEG-IFN/RBV lead-in therapy is performed during 0-4 weeks, then add boceprevir from week 5 (boceprevir+ PEG-IFN/RBV). If HCV RNA is undetectable during 8-24 weeks, boceprevir+PEG-IFN/RBV triple therapy will be administered from week 5 to week 32.
- Patients With 48 Weeks Therapy: For non-cirrhotic patients whose response of previous HCV therapy with PEG-IFN/RBV were relapse or partial response, PEG-IFN/RBV lead-in therapy is performed during 0-4 weeks, then add boceprevir from week 5 (boceprevir+ PEG-IFN/RBV). If HCV RNA is detectable at week 8 and undetectable at week 24, boceprevir+ PEG-IFN/RBV triple therapy will be administered from week 5 to week 32, followed by additional 12 weeks of PEG-IFN/RBV therapy.
- Null Responder or Cirrhotic Patients: For null responder or cirrhotic patients, PEG-IFN/RBV lead-in therapy is performed during 0-4 weeks, then add boceprevir from week 5 to 48.
Period: Overall Study
Arm/Group | Patients With 32 Week Therapy | Patients With 48 Weeks Therapy | Null Responder or Cirrhotic Patients
Started | 4 | 0 | 8
Completed | 4 | 0 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Twelve patients was enrolled. Patients with 32 week therapy are belong to arm A, and all patients were 20 years or older; HCV GT1/HBV dual infections; history of refractory to prior PEG-IFN/RBV treatment for at least 12 weeks; compensated liver disease consistent with chronic hepatitis C and/or B, without other etiology
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With 32 Week Therapy | Patients With 48 Weeks Therapy | Null Responder or Cirrhotic Patients | Total
Number analyzed (Participants) | 4 | 0 | 8 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (16.0) |  | 50.6 (9.2) | 48.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 4 | 4
  Male | 4 |  | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Full Analysis Set Participants Who Received HCV Anti-viral Therapy With Sustained Virological Response (SVR)
Description: The methods used to assess this outcome measure is by full-analysis set (FAS), which is defined as undetectable HCV-RNA at follow-up Week 24 in subjects receiving ≥1 dose of any antiviral medication (Boceprevir/peginterferon/ribavirin)
Time Frame: week 24
Population: For survey the total 12 chronic hepatitis C patients by FAS in different arms in this clinical- trial.
  Outcome Measure Data Table: For survey the total 8 chronic hepatitis C patients had SVR by FAS in different arms in this clinical- trial.
Measure: Number; unit: participants
Groups:
- Null Responder or Cirrhotic Patients: For null responder or cirrhotic patients, PEG-IFN/RBV lead-in therapy is performed during 0-4 weeks, then add boceprevir from week 5 to 48.
  Stop trial intervention for boceprevir, PEG-IFN and RBV: Stop trial intervention for patients with 32 week therapy (arm A): for all patients, if HCV RNA is more than 100 IU/ml at week 12 or HCV RNA is detectable at week 24, therapy will be stopped.
  Stop trial intervention for patients with 48 weeks therapy (arm B): for all patients, if HCV RNA is more than 100 IU/ml at week 12 or HCV RNA is detectable at week 24, therapy will be stopped.
  Stop trial intervention for for null responder or cirrhotic patients: (arm C) for all patients, if HCV RNA is more than 100 IU/ml at week 12 or HCV RNA is detectable at week 24, therapy will be stopped.
Arm/Group | Patients With 32 Week Therapy | Patients With 48 Weeks Therapy | Null Responder or Cirrhotic Patients
Number analyzed (Participants) | 4 | 0 | 8
participants | 4 |  | 4
Statistical Analysis 1: Comparison: Patients With 32 Week Therapy vs Patients With 48 Weeks Therapy vs Null Responder or Cirrhotic Patients; Test type: Other — The evaluation of SVR rate was based on full-analysis-set (FAS) and modified intention-to-treat population (mITT). FAS population included subjects receiving ≥ 1 dose of any antiviral agents (boceprevir and/or PEG-IFN, and/or RBV). MITT population included subjects receiving ≥ 1 dose of boceprevir; p = 0.01, Chi-squared

2. Secondary Outcome: Key Secondary Endpoint of This Clinical Trial-SVR in mITT
Description: The total 7 patients had SVR by mITT in this clincial-trial, which is defined as undetectable HCV-RNA at follow-up Week 24 in subjects receiving ≥1 dose of Boceprevir
Time Frame: week 24
Population: MITT population included subjects receiving ≥ 1 dose of boceprevir.
Measure: Number; unit: participants
Arm/Group | Patients With 32 Week Therapy | Patients With 48 Weeks Therapy | Null Responder or Cirrhotic Patients
Number analyzed (Participants) | 4 | 0 | 7
participants | 4 |  | 3

3. Other Pre Specified Outcome: The Other Responses in the mITT Population/Safty- HBV Virologic Response
Description: HBV virologic response, defined as serum HBV DNA levels to < 200 IU/mL at follow-up week 24 among patients with detectable HBV DNA at baseline
Time Frame: week 24
Measure: Number; unit: participants
Arm/Group | Patients With 32 Week Therapy | Patients With 48 Weeks Therapy | Null Responder or Cirrhotic Patients
Number analyzed (Participants) | 4 | 0 | 8
participants | 0 |  | 0

ADVERSE EVENTS:
Time Frame: The specific period of time over which adverse event data were collected from baseline to end of follow up.
Description: Adverse events (AEs) data were collected on all patients during their treatment and posttreatment 6-month follow-up period. These data included clinical and laboratory grade 3 or 4 AEs, serious adverse events (SAEs), and special interest events, such as grade 2 or higher anemia events, infections, hepatic decompensation and other cytopenias.
Arm/Group | Patients With 32 Week Therapy | Patients With 48 Weeks Therapy | Null Responder or Cirrhotic Patients
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0 | 1/8
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With 32 Week Therapy (N=4) | Patients With 48 Weeks Therapy (N=0) | Null Responder or Cirrhotic Patients (N=8)
pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 — pregnancy
Fever (Infections and infestations) | 0 | 0 | 0 — Fever due to suspect infection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With 32 Week Therapy (N=4) | Patients With 48 Weeks Therapy (N=0) | Null Responder or Cirrhotic Patients (N=8)
Gastroenterology (Gastrointestinal disorders) | 4 | 0 | 8 — The most frequent AEs during therapy course were gastroenterological (12 subjects, 100%)
Dermatology (Skin and subcutaneous tissue disorders) | 3 | 0 | 7 — The most frequent AEs during therapy course was dermatologic (10 subjects, 83.3%) manifestations

LIMITATIONS AND CAVEATS:
The limitation of this study is the limited case number.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No